CLINICAL TRIAL: NCT02541149
Title: Evaluation of Annexin A2 as a Novel Diagnostic Marker for Hepatocellular Carcinoma in Egyptian Patients
Brief Title: Annexin A2 as a Novel Diagnostic Marker in Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: Annexin A2
Record Dates: First submitted 2015-09-01; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1:: Fifty patients with early stage hepatocellular carcinoma(BCLC stage A)
  Interventions: Procedure: blood sample
- Group 2: Twenty five patients with chronic liver disease diagnosed based on clinical, laboratory, and ultrasonographic investigations;
  Interventions: Procedure: blood sample
- Group 3: Control Group: Fifteen healthy, age and sex-matched subjects with seronegative hepatitis viral markers
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample

SUMMARY:
This study aimed to investigate the clinical utility of Annexin A2 serum level as a novel diagnostic marker of hepatocellular carcinoma (HCC) and to correlate its level with alpha fetoprotein the current marker ofhepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This study was carried out in HCC clinic , Ain Shams University Hospitals, Cairo; Egypt and included :Group 1: Fifty patients with early stage hepatocellular carcinoma(BCLC stage A); Group 2:Twenty five patients with chronic liver disease diagnosed based on clinical, laboratory, and ultrasonographic investigations; Control Group: Fifteen healthy, age and sex-matched subjects with seronegative hepatitis viral markers .All groups were subjected to thorough history taking, full clinical examination, and laboratory investigations including viral hepatitis markers: HBsAg and HCV antibodies using ELISA technique and HCV RNA using real time PCR for HCV antibody positive patients, AFP by electrochemiluminescence and Annexin A2 estimation using ELISA technique.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for HCC cases:

  1. Confirmed diagnosis of HCC according to the European association of study of liver diseases [13].
  2. Early stage HCC (Stage A), using the Barcelona Clinic Liver Cancer (BCLC) staging system, (single or 3 nodules < 3cm PS 0) For all participants:.
* Informed consent from all participants before enrollment in the study.

Exclusion Criteria:

* For HCC patients:

  1-Imtermediate or advanced stage HCC as defined by BCLC 2. Major vascular tumor invasion or metastasis confirmed by radiological imaging studies.

  3. Patients with other suspected solid malignancies or metastatic liver tumors, 4. Other types of chronic liver diseases (CLD) such as autoimmune hepatitis and primary biliary cirrhosis.
* For all participants:

  * Refusal to participate in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Egyptian patients attending outpatient clinic for HCC , Ain Shams University Hospitals, Cairo Egypt (Group 1&2)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
serum Annexin A2 in patients with hepatocellular carcinoma, chronic liver disease and healthy subjects | 1 month
  to determine the clinical utility of Annexin A2 serum level as a novel diagnostic marker of hepatocellular carcinoma (HCC) and to correlate its level with alpha fetoprotein the current marker of (HCC).